CLINICAL TRIAL: NCT03938701
Title: Near-infrared Fluorescence Molecular Imaging of Adalimumab-800CW to Elucidate the Drug Distribution Throughout Inflamed Tissue in Inflammatory Bowel Disease and Rheumotoid Arthritis
Brief Title: Fluorescence Imaging of IBD and RA Using Adalimumab-800CW
Acronym: STRATIFY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL75246.042.20
Record Dates: First submitted 2019-02-25; First posted 2019-05-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: IBD; Rheumatoid Arthritis
Keywords: Molecular imaging; Adalimumab-800CW; Fluorescence; Inflammatory bowel disease; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammatory Bowel Diseases | interventions — Adalimumab; Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1. Fluorescence imaging of inflammatory bowel disease and rheumatoid arthritis with adalimumab-800CW (Experimental): Fluorescence imaging with 4.5 mg adalimumab-800CW in inflammatory bowel disease and rheumatoid arthritis.
  Interventions: Drug: Adalimumab-800CW; Device: Fluorescence Imaging
- 2. Fluorescence imaging of inflammatory bowel disease and rheumatoid arthritis with adalimumab-800CW (Experimental): Fluorescence imaging with 15 mg adalimumab-800CW in inflammatory bowel disease and rheumatoid arthritis.
  Interventions: Drug: Adalimumab-800CW; Device: Fluorescence Imaging
- 3. Fluorescence imaging of inflammatory bowel disease and rheumatoid arthritis with adalimumab-800CW (Experimental): Fluorescence imaging with 25 mg adalimumab-800CW in inflammatory bowel disease and rheumatoid arthritis.
  Interventions: Drug: Adalimumab-800CW; Device: Fluorescence Imaging
- 4. Fluorescence imaging of inflammatory bowel disease and rheumatoid arthritis (Experimental): Fluorescence imaging without adalimumab-800CW in inflammatory bowel disease and rheumatoid arthritis.
  Interventions: Device: Fluorescence Imaging

INTERVENTIONS:
Drug: Adalimumab-800CW — Intravenous administration of 4.5 mg, 15 mg or 25 mg 2 - 4 days prior to the fluorescence imaging
  Other Names: Humira
  Arms: 1. Fluorescence imaging of inflammatory bowel disease and rheumatoid arthritis with adalimumab-800CW; 2. Fluorescence imaging of inflammatory bowel disease and rheumatoid arthritis with adalimumab-800CW; 3. Fluorescence imaging of inflammatory bowel disease and rheumatoid arthritis with adalimumab-800CW
Device: Fluorescence Imaging — Rheumatoid arthritis: a flexible fiber-bundle is attached to a fluorescence camera platform to enable the detection of fluorescence signals open-air by using a black-box.
  Inflammatory bowel disease: a flexible fiber-bundle is attached to a fluorescence camera platform to enable the detection of fluorescence signals. The fluorescence fibre-probe is inserted through the standard working channel of the standard clinical endoscope. Fluorescence imaging will be performed during standard clinical colonoscopy.
  Other Names: Quantified fluorescence molecular endoscopy

SUMMARY:
Inflammatory bowel disease (IBD) and rheumatoid arthritis (RA) are both auto-immune diseases that are characterized by chronic relapsing inflammation of respectively the ileocolonic tissue and the synovium. Pathogenesis of both auto-immune diseases is attributed to the proinflammatory cytokine tumor necrosis factor α (TNFa). Adalimumab is a human monoclonal anti-TNF antibody used for treating patients with moderate to severely active IBD and RA. However, current rates of therapeutic nonresponsiveness to this antibody are variable and difficult to predict in advance, whereas patients are potentially exposed to a non-effective treatment and its potential side effects; while clinical deterioration progresses. A key unmet need is the development of a predictive tool for assessment of a therapeutic (non-) response to patients and finding an optimal dose strategy in individual patients before initiating anti-TNF therapy. Unfortunately, we currently lack crucial information about drug distribution of the drug of interest throughout the targeted inflamed tissue itself. Therefore, it remains unknown in both IBD and RA, if the drug reaches its target (in sufficient amounts) and how local drug concentrations are related to therapeutic response. Thus, we linked adalimumab to a fluorescent dye (adalimumab-800CW) in order to create a fluorescent signal of the labelled drug in the diseased tissue that we can visualize and quantify with dedicated optical fluorescence imaging systems. We hypothesize that this tracer will bind to TNFa in the mucosa/synovium and thus create a map of medicine distribution in vivo due to colocalization of the fluorescent labelled compound. Therefore, the aim of this study is to assess the feasibility of fluorescent molecular imaging of adalimumab-800CW in IBD and RA patients.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion criteria:

* Established IBD or RD diagnosis
* Active disease.

  * IBD cohort: clinically active disease of the bowel defined either clinically as at least mild activity using dedicated scoring indices (for definitions of disease activity, see below) or biochemically active disease as defined by a faecal calprotectin > 200 µg/g;
  * RA cohort: clinically active disease of at least one joint of the hand as assessed by a rheumatologist;
* Age of 18 years or older and mentally competent;
* Written informed consent.

IBD patients must already have an ileocolonoscopy scheduled due to a clinical indication.

For female subjects which are of childbearing potential, are premenopausal with intact reproductive organs or are less than 2 years postmenopausal

* A negative pregnancy test must be available
* Willing to ensure that she uses effective contraception during the study and for 3 months thereafter.

Exclusion criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* A potential female subject that is pregnant or provides breastfeeding will be excluded from participation in this study.
* The exclusion criterium that is specific for RD patients involves a skin type above type 3 according to the Fitzpatrick scale due to feasibility of the MDSFR/SFF spectroscopy measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety: number of participants with symptoms or changes in vital signs (blood pressure, heart rate and temperature) that are related to administration of adalimumab-800CW | Up to 30 minutes after stop tracer injection
  To determine the safety of adalimumab-800CW in inflammatory bowel disease (IBD) and rheumatoid arthritis patients by monitoring of vital signs (blood pressure, heart rate and temperature) before, during and after tracer infusion.
  These vital signs are measured before tracer administration, directly after and then every 15 minutes until 1 hour after tracer administration.
Safety: number of participants with (serious) adverse events that are related to the administration of adalimumab-800CW | Up to 24 hours after tracer injection
  (serious) adverse events will be monitored until 24 hours after tracer administration.
Discrimination of inflamed and normal tissue based on in vivo fluorescence measurements from adalimumab-800CW gained during fluorescence imaging of the hand of rheumatoid arthritis patients | Up to 1 year
  The target-to-background/contrast-to-noise ratio will be calculated after fluorescence imaging. These results will be related to the gold standard clinical care to evaluate the feasibility of molecular fluorescence imaging using the tracer adalimumab-800CW for the evaluation of drug distribution in patients with rheumatoid arthritis.
Discrimination of inflamed and normal tissue based on in vivo and ex vivo fluorescence measurements from adalimumab-800CW gained during fluorescence endoscopy in patients with ulcerative colitis (UC). | Up to 1 year
  The target-to-background/contrast-to-noise ratio will be calculated after fluorescence molecular endoscopy (FME) and MDSFR/SFF spectroscopy. These results will be related to the gold standard clinical care to evaluate the feasibility of fluorescence molecular endoscopy using the tracer adalimumab-800CW for the evaluation of drug distribution in patients with ulcerative colitis.
Discrimination of inflamed and normal tissue based on in vivo and ex vivo fluorescence measurements from adalimumab-800CW gained during fluorescence endoscopy in patients with Crohn's disease (CD). | Up to 1 year
  The target-to-background/contrast-to-noise ratio will be calculated after fluorescence molecular endoscopy (FME) and MDSFR/SFF spectroscopy. These results will be related to the gold standard clinical care to evaluate the feasibility of fluorescence molecular endoscopy using the tracer adalimumab-800CW for the evaluation of drug distribution in patients with Crohn's disease.

SECONDARY OUTCOMES:
The correlation between the fluorescence intensity and the disease activity measured with the DAS28 in patients with RA. | Up to 1 year
  The DAS28 (Disease Activity Score 28) is developed and validated by the EULAR (European League Against Rheumatism) to measure the progress and improvement of Rheumatoid Arthritis by measuring 28 joints. When looking at these joints, both the number of joints with tenderness upon touching and swelling are counted. Furthermore, the erythrocyte sedimentation rate is measured and a patients assessment of disease activity during the preceding 7 days is measured on a scale between 0 and 100, where 0 is 'no activity' and 100 is 'highest activity possible'.
  DAS28 values range from 0.49 to 9.07 while higher values mean a higher disease activity. A DAS28 below the value of 2.6 is interpreted as Remission. Between 2.6 and 3.2 as low disease activity, and between 3.2 and 5.1 as moderate. Above 5.1 is indicated as high disease activity.
Calculation of optical properties with MDSFR/SFF spectroscopy in patients with RA | Up to 1 year
  To quantify the optical properties, in vivo using multi-diameter single-fiber reflectance, single-fiber fluorescence (MDSFR/SFF) spectroscopy measurements;
The correlation between fluorescence intensity and the clinical disease activity score in ulcerative colitis using the SCCAI; | Up to 1 year
  The SCCAI is a diagnostic questionnaire to assess the severity of symptoms in patients with ulcerative colitis. The score ranges from 0 to 19 based on questions on topics regarding the bowel frequency, urgency of defecation, blood in stool and general health. A score of 5 or higher indicates active disease.
The correlation between fluorescence intensity and the endoscopic disease activity score in ulcerative colitis using the Mayo endoscopic subscore; | Up to 1 year
  The endoscopic Mayo Score (Mayo endoscopic subscore) evaluates ulcerative colitis stage, based only on endoscopic exploration. Endoscopic activity is based upon the assessment of a few features, such as the presence of erythema, visibility of the vascular pattern, friability, erosions, spontaneous bleeding and (large) ulcerations. Each score indicates endoscopic activity: 0 = inactive disease tot 3 = severely active disease.
  3-5 = mild activity 6-10 = moderate activity >10 = severe activity
The correlation between fluorescence intensity and the clinical disease activity score in Crohn's disease using the Crohn's Disease Activity Index (CDAI). | Up to 1 year
  The CDAI quantifies the symptoms of patients with CD. The index consists of 8 factors, each summed after adjustment with a weighting factor. Symptoms are scored over the last 7 days and include: number of soft/liquid stools, general well being, severity of abdominal pain, number of complications, ant-diarrhea drug use, abdominal mass, hematocrit, body weight.
  Remission is defined as CDAI < 150 and severe disease as CDAI > 450.
The correlation between fluorescence intensity and the disease activity score in Crohn's disease using the SES-CD score | Up to 1 year
  SES-CD (Simple Endoscopic Score for Crohn Disease) is a endoscopic assessment tool for patients with Crohn's disease. Four parameters are evaluated: ulcers, surface involved by disease, surface involved by ulcerations and narrowings.
  0-2 = remission 3-6 = mild endoscopic activity 7-15 = moderate endoscopic activity >15 = severe endoscopic activity
The correlation and validation of fluorescence signals detected in vivo to the pathology of biopsies for IBD patients; | Up to 1 year
  Pathology findings are correlated to fluorescence signals to determine if pathology results (inflammation) correspond to fluorescence signals (high fluorescence) and vice versa, normal tissue corresponds too low fluorescence signals.
Quantification of fluorescence signals in vivo and ex vivo of inflamed and normal tissue using multi-diameter single-fiber reflectance, single-fiber fluorescence (MDSFR/SFF) spectroscopy measurements in IBD patients; | Up to 1 year
  The measurements with MDSFR/SFF are performed on the same tissue: in vivo during endoscopy and ex vivo on the biopsies. Therefore they are considered as one measurement outcome.
  Measurements are taken from both normal tissue and inflammation tissue.
Correlation in IBD between the detected fluorescence signals in vivo and the clinical response to induction therapy at week 14. | Up to 1 year
  Values of clinical disease activity scores (SCCAI for UC and CDAI for CD) will be obtained at week 14 from the patient's electronic medical chart in order to determine the correlation with the target-to-background ratio measured at baseline during fluorescence molecular endoscopy (FME) and MDSFR/SFF spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter B. Nagengast, MD, PhD, PharmD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No